CLINICAL TRIAL: NCT00242515
Title: Preemptive CD8+ T-cell Depleted Donor Lymphocyte Infusion (DLI) Following Nonmyeloablative Stem Cell Transplantation (NMT) for Acute Myeloid Leukemia (AML) or High Risk Myelodysplastic Syndrome (MDS)
Brief Title: T-cell Depleted Donor Lymphocyte Infusion (DLI)for Acute Myeloid Leukemia (AML) or High Risk Myelodysplastic Syndrome (MDS)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP02/28/04
Record Dates: First submitted 2005-10-19; First posted 2005-10-20 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: High risk Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

INTERVENTIONS:
Procedure: CD8+ T-cell depleted donor lymphocyte infusion

SUMMARY:
Primary Objectives:

This a pilot project to determine the feasibility of the preemptive CD8+ depleted T-cell donor lymphocyte infusion (DLI) in:

* Reducing the incidence of graft versus host disease (GVHD) based on standard classification of acute and chronic GVHD
* Improving hte disease remission rate in comparison with our previous study results.

Secondary Objectives:

* To investigate the impact of CD8+ depleted T-cell DLI in hematopoietic chimerism, and immunologic recovery of transplant patients.

DETAILED DESCRIPTION:
The scientific investigation in this study protocol:

1. Define the role of preemptive and specific DLI in preserving the GVL effect in the setting of NMT. The ability of selecting components of T cells for transplant and DLI will allow us to test the hypothesis of distinctive roles in subsets of T cells. It was found that CD8-depleted DLI was administered to prevent relapse after TCD (T-cell depleted) BMT (bone marrow as the stem cell source) or CD34-selected PBSC.

   Whether preemptive CD8-depleted DLI can perform this function after nonmyeloablative transplantation (NMT) needs to be established, as proposed in our study. If there turns out to be a role for DLI in these circumstances, a CD8-depleted lymphocyte product that can limit GVHD would be a very attractive option. We would also define the relationship of the level of donor chimerism and disease control.
2. Investigate the impact of CD8-depleted DLI in NMT at specific doses and time points for the reduction of GVHD. The GVHD pattern may vary between different ethnic populations as suggested by our earlier NMT study. Our current proposed study will further shed light on the optimal GVHD prophylaxis regimen in the Singapore patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of AML or high risk MDS in the following disease stages: Induction failure, first or subsequent remission, or untreated first relapse.
2. Patient must have an HLA-compatible donor willing and capable of donating peripheral blood stem cells preferably or bone marrow progenitor cells using conventional techniques, and lymphocytes if indicated (HLA-compatible defined as 5/6 or 6/6 matched related or 6/6 molecular matched unrelated donor)
3. Both patient and donor must sign written informed consent forms.
4. Patients must have:

   * ECOG PS </= 2;
   * Ejective fraction > 40%;
   * DLCO > 40% of predicted;
   * Serum bilirubin </= 1.5x institutional upper limit of normal;
   * SGPT (ALT) and SGOT (AST) </= 2.5x institutional upper limit of normal;
   * Serum creatinine </= 2x upper limit of normal;
   * Creatinine clearance >/= 60mL/min. However, renal dysfunction is not an absolute contraindication for NMT as dialysis can be performed during NMT.

Exclusion Criteria:

1. Not fulfilling any of the inclusion criteria
2. Active life-threatening infection
3. Overt untreated infection
4. HIV positivity, hepatitis B or C antigen positivity with active hepatitis
5. Pregnant or lactating women
6. Donor contraindication (HIV seropositive confirmed by Western blot; hepatitis B antigenemia)
7. Unable to donate bone marrow or peripheral blood due to concurrent medical condition

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2005-03; Study Completion 2008-03

PRIMARY OUTCOMES:
Incidence rate of acute and chronic GVHD
Disease remission rate post CD8+ depleted T-cell DLI

SECONDARY OUTCOMES:
Hematopoietic chimerism and immunologic recovery post CD8+ depleted T-cell DLI

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Shing Chen, MD, Principal Investigator — National University Hospital/National University Singapore
Locations (1):
- Department of Hematology-Oncology, National University Hospital, Singapore, Singapore